CLINICAL TRIAL: NCT04423133
Title: Bilingual Family Literacy Program Pilot: Ready and Healthy for Kindergarten
Brief Title: Bilingual Family Literacy Program Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Manuel E. Jimenez, MD, MS, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro2020000656
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Language Development; Literacy; Health Behavior
Keywords: Language development; Health routines; Literacy
MeSH Terms: conditions — Literacy; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online Family Literacy Program (Experimental): The Ready and Healthy for Kindergarten program is a bilingual family literacy program that uses anticipatory guidance on health routines (e.g., physical activity) to introduce language and literacy skills to children and their families delivered via an online video conference format.
  Interventions: Behavioral: Online Family Literacy Program

INTERVENTIONS:
Behavioral: Online Family Literacy Program — Parent-child dyads will participate in 8 weekly online health-themed workshops that introduce language and literacy skills. Participants will also receive 2-3 text messages per week for the duration of the program and children's books.

SUMMARY:
This study will examine the feasibility of implementing a virtual bilingual health-focused family literacy program.

DETAILED DESCRIPTION:
"Ready and Healthy for Kindergarten" is a bilingual family literacy program that uses anticipatory guidance on important health routines to introduce critical language and literacy skills to young Latino children entering Kindergarten and their families.

The objectives of this study are 1) To assess the feasibility of implementing the bilingual family literacy program online via video conference by collecting information on family attendance and participation, 2) To examine the acceptability of the program, and 3) To explore preliminary effects of the program on the family health and language routines as well as child language and literacy skill acquisition.

ELIGIBILITY:
Inclusion Criteria:

* Preferred language either Spanish or bilingual (English and Spanish)
* Parent or legal guardian of the child
* Parent Age ≥ 18

Exclusion Criteria:

* Children not entering Kindergarten.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Number of sessions attended by participants | 8 weeks
  Data on the number of sessions attended by participants will be used to assess the feasibility of the online family literacy program.
Acceptability of the program | 8 weeks
  Data on acceptability of the program will be collected via parent surveys

SECONDARY OUTCOMES:
StimQ Reading Scale | Baseline, 8 weeks
  Reading activity will be measured using the StimQ Reading Scale. The StimQ is a structured interview. Individual items are summed and scores range from 0 to 19. Higher scores reflect higher reading activities.
StimQ Parental Verbal Responsivity Scale | Baseline, 8 weeks
  Parent verbal responsiveness will be measured using the StimQ Parental Verbal Responsivity Scale. The StimQ is a structured interview. Individual items are summed and scores range from 0 to 7. Higher scores reflect higher parent verbal responsiveness.
Child Literacy Skills | Baseline, 8 weeks
  Investigator developed assessments of child alphabet knowledge and sight word recognition. Higher scores reflect higher literacy skills.
Family Health Routines Assessment | Baseline, 8 weeks
  Descriptive survey measuring family health routines and behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel E Jimenez, MD, MS, Principal Investigator — Rutgers Biomedical Health Sciences
Locations (1):
- Child Health Institute of NJ, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No